CLINICAL TRIAL: NCT05141968
Title: The Effects of Vitamin D Supplementation on Glycemic Control in Children With Type 1 Diabetes Mellitus in Gaza Strip, A Randomized Controlled Trial
Brief Title: Vitamin D Supplementation and Glycemic Control Improvement Among Type 1 Diabetic Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Principal Investigator Heba Mohammed Arafat, Department of Chemical Pathology, School of Medical Sciences, Health Campus, Universiti Sains Malaysia, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: AlAzharDiabetes
Record Dates: First submitted 2021-10-30; First posted 2021-12-02 (Actual); Last update posted 2021-12-02 (Actual); Status verified 2021-11

CONDITIONS: Type 1 Diabetes Mellitus; Vitamin D Deficiency
Keywords: Vitamin D Supplementation; Glycemic Control; Type 1 Diabetes Mellitus; Gaza Strip; Randomized Controlled Trial.
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Vitamin D Deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin D supplements group (Experimental): Group A: is the interventional group that supplemented with vitamin D tablets contain 2000 IU once time daily with a meal, for 3 months of intervention.
  Interventions: Dietary Supplement: vitamin D supplements (2000 IU/day)
- Control group (No Intervention): Group B: is the control group, that did not receive any supplements.

INTERVENTIONS:
Dietary Supplement: vitamin D supplements (2000 IU/day) — The interventional (experimental) group received vitamin D supplements (2000 IU/day). According to previous studies and after the direct supervision from the treating pediatrician and endocrinologist, the best preparation and dosage of vitamin D was used (According to FDA the recommended dose for children age 1 year and older is 2,000 IU/day).
  Arms: Vitamin D supplements group

SUMMARY:
Type 1 diabetes mellitus (T1DM) is an immune-mediated disease characterized by diminished insulin secretion due to damage to islets of Langerhans in the pancreas, which eventually results in high levels of glucose in the blood. According to World Diabetes Foundation, in Palestine, 4.4% of diabetic patients are diagnosed with T1DM, while 95.3% are diagnosed with type 2 diabetes (T2DM) (World Diabetes Foundation, 2020).

Observational studies have reliably provided evidence that T1DM patients with acceptable glycemic control have higher 25(OH)D levels than T1DM with lesser glycemic control. Additionally, it has been specified by some of the research-based studies that there is a strong connection between the deficiency of vitamin D and the incidence of T1DM.

In interventional studies of T1DM children and adults, repletion of vitamin D in deficient individuals improved HbA1c in a period of 12 weeks. Participants were more likely to achieve HbA1c < 7.8% if they had higher 25(OH)D levels on week 12 than on baseline, especially if 25(OH)D levels were exceeded 51 nmol/l.

According to the Food and Drug Administration (FDA), The Institute of Medicine's (IOM) recommended Upper Limit (UL) for chronic Vitamin D intake for infants (children less than 1 year of age) is 25 mcg/day (1,000 IU/d), and for children age 1 year and older the recommended UL is 50 mcg/day (2,000 IU/d) (Institute of Medicine Standing Committee on the Scientific Evaluation of Dietary Reference Intakes, 1997).

Despite a large amount of evidence from observational and experimental studies supporting the effects of vitamin D on glucose metabolism and the immune system, results from clinical studies remain inconsistent, which makes it impossible to recommend vitamin D supplementation for the treatment of T1DM. Therefore, this study aimed to investigate the status of vitamin D among T1DM children for vitamin and to examine the effects of vitamin D supplementation on glycemic control in children with T1DM. This is the first randomized controlled trial that studied the effects of vitamin D supplementation on glycemic control among T1DM children in the Gaza Strip, Palestine.

DETAILED DESCRIPTION:
2.1 Study design The study design was experimental, A randomized controlled trial. 2.2 Study setting The study was conducted at the endocrinology outpatients' clinic at AL-RANTISI PEDIATRIC HOSPITAL in Gaza Strip.

2.3 Study Sample After getting the ethical approval, data were collected throughout 3 months, starting from October 2017 to January 2018. In this period, 80 children who were less than 14 years old were diagnosed with T1DM which was indicated through fasting blood glucose level greater than 126 mg/dl or HbA1c cut point of ≥6.5% (American Diabetes Association, 2010), and had vitamin D deficiency which indicated by its levels of less than 12 ng/ml (Sullivan, 2019), were recruited from endocrinology outpatients' clinic at AL-RANTISI PEDIATRIC HOSPITAL in Gaza Strip.

2.4 Sampling

A stratified random sampling technique was applied to assign children with the previously mentioned criteria into two groups. The first group is the interventional (experimental) group that received vitamin D supplements (2000 IU/day) and the second group is the control group that did not receive any supplements. Both groups were on their regular diet and treatment, but one group was put on vitamin D supplement and the other group received a placebo instead. According to previous studies and after the direct supervision from the treating pediatrician and endocrinologist, the best preparation and dosage of vitamin D was used (According to FDA the recommended dose for children age 1 year and older is 2,000 IU/day). The two groups were defined as follows:

Group A: is the control group, that received a placebo as a supplement. Group B: is the interventional group that supplemented with vitamin D tablets containing 2000 IU once time daily with a meal, for 3 months of intervention.

Concerning the laboratory investigations; vitamin D status was assessed by measuring the concentration of 25-hydroxyvitamin D (25(OH)D) in the children's serum. Levels of 25(OH)D were interpreted as deficiency (≤20 ng/ml or ≤50 nmol/L), insufficiency (21-29 ng/ml or 52.5-72.5 nmol/L), and sufficiency (30-100 ng/ml ng/ml or 75-250 nmol/L). The glycated hemoglobin levels are defined based on the control of diabetes, as good control (HbA1c<7.8%), moderate control (HbA1c:7.8%-9.9%), and poor control (HbA1c>9.9%).

2.5 Tools of Data Collection

Children's health assessment structure interview sheet was used to collect data. It was constructed by the researchers based upon relevant literature. The questionnaire consisted of three parts:

Part I: Children's socio-demographic characteristics This part was aimed to collect socio-demographic characteristics for both interventions, and control groups before the intervention such as age, gender, number of family members, and level of education.

Part II: Children's current health history It covered the history of the discovery of diabetes, duration of diabetes, type of insulin, family history of diabetes, and periodic test for diabetes. This part had been used before the intervention for both the intervention and control groups.

Part III: Children's laboratory investigations This part addressed HbA1c that was investigated and recorded before and after the interference for both interventions, and control groups. Additionally, vitamin D status was assessed and recorded before the intervention for both interventions, and control groups.

2.6 Statistical analysis Data was entered and statistically analyzed using a statistical package for social sciences (SPSS) version 26 database for windows 10. Descriptive statistics were used to summarize the socio-demographic characteristics of subjects. Numerical data like 25-(OH)D levels, and HbA1c, were presented as mean (SD) or median (IQR) based on their normality distribution. Categorical data were presented as frequency (percentage). The chi-square test was used for categorical data comparison. Analysis of quantitative data between two groups was done using unpaired t-test. Pearson correlation coefficients between continuous variables were used as a measure of association. A p-value <0.05 was considered statistically significant.

ELIGIBILITY:
The eligibility criteria are:

Criteria for children with T1DM:

Inclusion criteria for children with T1DM:

* Children (4-14 years of age) of both genders, with a T1DM.
* Not on vitamin D Supplementation. Exclusion criteria for children with T1DM
* Age ≤ 4 or more than14 years old
* Patients with T2DM
* Children had received vitamin D supplements

Ages: 4 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2021-06-16 (Actual)

PRIMARY OUTCOMES:
Percent of HbA1c in children with T1DM for both intervention, and control groups. | Three Months
  Change of glycemic control in children with T1DM. The glycohemoglobin levels are defined based on the control of diabetes, as good control (HbA1c<7.8%), moderate control (HbA1c:7.8%-9.9%), and poor control (HbA1c>9.9%). The percent of HbA1c was measured and recorded before and after the interference for both interventions, and control groups, (the interventional group was supplemented with vitamin D tablets containing 2000 IU once time daily with a meal, for 3 months of intervention).
  Children's health assessment structure interview sheet was used to collect data. It was constructed by the researchers based upon relevant literature. The questionnaire consisted of three parts Part I: Children's socio-demographic characteristics Part II: Children's current health history Part III: Children's laboratory investigations

SECONDARY OUTCOMES:
Concentration of Vitamin D for both intervention, and control groups | Three Months
  Screening for vitamin D deficiency among type 1 diabetic children. The vitamin D status was assessed by measuring the concentration of 25-hydroxyvitamin D (25(OH)D) in the children's serum. Levels of 25(OH)D were interpreted as deficiency (≤20 ng/ml or ≤50 nmol/L), insufficiency (21-29 ng/ml or 52.5-72.5 nmol/L), and sufficiency (30-100 ng/ml ng/ml or 75-250 nmol/L). Vitamin D status was assessed and recorded before and after the intervention for both interventions, and control groups.

CONTACTS AND LOCATIONS:
Overall Officials: Heba A Al Sarraj, PhD, Study Chair — Department of Laboratory Medicine, Al Azhar University-Gaza, Gaza Strip, Palestine; Ashraf J Shaqaliah, Master, Study Director — Department of Laboratory Medicine, Al Azhar University-Gaza, Gaza Strip, Palestine; Heba M Arafat, PhD, Principal Investigator — Department of Chemical Pathology, School of Medical Sciences, Universiti Sains Malaysia; Ohood M Shamallakh, Master, Principal Investigator — Department of a Medical Laboratory Sciences, Faculty of Health Sciences, Islamic University of Gaza; Kholoud M Shamallakh, Master, Principal Investigator — Department of a Medical Laboratory Sciences, Faculty of Health Sciences, Islamic University of Gaza
Locations (1):
- Al-Rantisi pediatric hospital, Gaza, Palestinian Territories

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Al-Agha, A. E., & Ahmad, I. A. (2015). Association among vitamin D deficiency, type 1 diabetes mellitus, and glycemic control. J Diabetes Metab, 6(594), 2.
- [Background] Aljabri KS, Bokhari SA, Khan MJ. Glycemic changes after vitamin D supplementation in patients with type 1 diabetes mellitus and vitamin D deficiency. Ann Saudi Med. 2010 Nov-Dec;30(6):454-8. doi: 10.4103/0256-4947.72265. PMID 21060157
- [Background] American Diabetes Association. Diagnosis and classification of diabetes mellitus. Diabetes Care. 2010 Jan;33 Suppl 1(Suppl 1):S62-9. doi: 10.2337/dc10-S062. No abstract available. PMID 20042775
- [Background] Bizzarri C, Pitocco D, Napoli N, Di Stasio E, Maggi D, Manfrini S, Suraci C, Cavallo MG, Cappa M, Ghirlanda G, Pozzilli P; IMDIAB Group. No protective effect of calcitriol on beta-cell function in recent-onset type 1 diabetes: the IMDIAB XIII trial. Diabetes Care. 2010 Sep;33(9):1962-3. doi: 10.2337/dc10-0814. PMID 20805274
- [Background] Busta, A., Alfonso, B., & Poretsky, L. (2011). Role of vitamin D in the pathogenesis and therapy of type 1 diabetes mellitus. In Type 1 diabetes-complications, pathogenesis, and alternative treatments (pp. 95-118): Intech, Rijeka.
- [Background] El-Sayed, R. E.-S. H., Abd El Raaouf, S. E. H., & Laimon, W. (2019). Effect of Vitamin D Supplementation on Glycemic Control in Children with Type 1 Diabetes Mellitus: A Randomized Clinical Trial. American Journal of Nursing, 7(4), 534-541.
- [Background] Elhamalawi, I. M. F. (2015). Assessment of serum Vitamin D in Type 1 Diabetic Patients from Gaza Strip.
- [Background] Gabbay MA, Sato MN, Finazzo C, Duarte AJ, Dib SA. Effect of cholecalciferol as adjunctive therapy with insulin on protective immunologic profile and decline of residual beta-cell function in new-onset type 1 diabetes mellitus. Arch Pediatr Adolesc Med. 2012 Jul 1;166(7):601-7. doi: 10.1001/archpediatrics.2012.164. PMID 22751874
- [Background] George PS, Pearson ER, Witham MD. Effect of vitamin D supplementation on glycaemic control and insulin resistance: a systematic review and meta-analysis. Diabet Med. 2012 Aug;29(8):e142-50. doi: 10.1111/j.1464-5491.2012.03672.x. PMID 22486204
- [Background] Griz LH, Bandeira F, Gabbay MA, Dib SA, Carvalho EF. Vitamin D and diabetes mellitus: an update 2013. Arq Bras Endocrinol Metabol. 2014 Feb;58(1):1-8. doi: 10.1590/0004-2730000002535. PMID 24728158
- [Background] Hafez M, Hassan M, Musa N, Abdel Atty S, Azim SA. Vitamin D status in Egyptian children with type 1 diabetes and the role of vitamin D replacement in glycemic control. J Pediatr Endocrinol Metab. 2017 Apr 1;30(4):389-394. doi: 10.1515/jpem-2016-0292. PMID 27997353
- [Background] Holick MF, Binkley NC, Bischoff-Ferrari HA, Gordon CM, Hanley DA, Heaney RP, Murad MH, Weaver CM; Endocrine Society. Evaluation, treatment, and prevention of vitamin D deficiency: an Endocrine Society clinical practice guideline. J Clin Endocrinol Metab. 2011 Jul;96(7):1911-30. doi: 10.1210/jc.2011-0385. Epub 2011 Jun 6. PMID 21646368
- [Background] nstitute of Medicine Standing Committee on the Scientific Evaluation of Dietary Reference Intakes. (1997). Dietary reference intakes for calcium, phosphorus, magnesium, vitamin D, and fluoride.
- [Background] Katsarou A, Gudbjornsdottir S, Rawshani A, Dabelea D, Bonifacio E, Anderson BJ, Jacobsen LM, Schatz DA, Lernmark A. Type 1 diabetes mellitus. Nat Rev Dis Primers. 2017 Mar 30;3:17016. doi: 10.1038/nrdp.2017.16. PMID 28358037
- [Background] Lamichhane AP, Crandell JL, Jaacks LM, Couch SC, Lawrence JM, Mayer-Davis EJ. Longitudinal associations of nutritional factors with glycated hemoglobin in youth with type 1 diabetes: the SEARCH Nutrition Ancillary Study. Am J Clin Nutr. 2015 Jun;101(6):1278-85. doi: 10.3945/ajcn.114.103747. Epub 2015 May 6. PMID 25948670
- [Background] Mitri J, Pittas AG. Vitamin D and diabetes. Endocrinol Metab Clin North Am. 2014 Mar;43(1):205-32. doi: 10.1016/j.ecl.2013.09.010. Epub 2013 Dec 12. PMID 24582099
- [Background] Mohammadian S, Fatahi N, Zaeri H, Vakili MA. Effect of vitamin d3 supplement in glycemic control of pediatrics with type 1 diabetes mellitus and vitamin d deficiency. J Clin Diagn Res. 2015 Mar;9(3):SC05-7. doi: 10.7860/JCDR/2015/10053.5683. Epub 2015 Mar 1. PMID 25954674
- [Background] Nwosu BU, Maranda L. The effects of vitamin D supplementation on hepatic dysfunction, vitamin D status, and glycemic control in children and adolescents with vitamin D deficiency and either type 1 or type 2 diabetes mellitus. PLoS One. 2014 Jun 11;9(6):e99646. doi: 10.1371/journal.pone.0099646. eCollection 2014. PMID 24918447
- [Background] Savastio S, Cadario F, Genoni G, Bellomo G, Bagnati M, Secco G, Picchi R, Giglione E, Bona G. Vitamin D Deficiency and Glycemic Status in Children and Adolescents with Type 1 Diabetes Mellitus. PLoS One. 2016 Sep 8;11(9):e0162554. doi: 10.1371/journal.pone.0162554. eCollection 2016. PMID 27607348
- [Background] Shih EM, Mittelman S, Pitukcheewanont P, Azen CG, Monzavi R. Effects of vitamin D repletion on glycemic control and inflammatory cytokines in adolescents with type 1 diabetes. Pediatr Diabetes. 2016 Feb;17(1):36-43. doi: 10.1111/pedi.12238. Epub 2014 Dec 18. PMID 25524404
- [Background] Sullivan, D. S., E. (2019). 25-Hydroxy Vitamin D Test. 2017(11/10). Retrieved from https://www.healthline.com/health/25-hydroxy-vitamin-d-test
- [Background] Walter M, Kaupper T, Adler K, Foersch J, Bonifacio E, Ziegler AG. No effect of the 1alpha,25-dihydroxyvitamin D3 on beta-cell residual function and insulin requirement in adults with new-onset type 1 diabetes. Diabetes Care. 2010 Jul;33(7):1443-8. doi: 10.2337/dc09-2297. Epub 2010 Mar 31. PMID 20357369
- [Background] World Diabetes Foundation. (2020). Palestine National Diabetes Program, WDF15-1304. Retrieved from https://www.worlddiabetesfoundation.org/projects/west-bank-and-gaza-wdf15-1304
- [Result] Al Sawah S, Compher CW, Hanlon AL, Lipman TH. 25-Hydroxyvitamin D and glycemic control: A cross-sectional study of children and adolescents with type 1 diabetes. Diabetes Res Clin Pract. 2016 May;115:54-9. doi: 10.1016/j.diabres.2016.03.002. Epub 2016 Mar 12. PMID 27242123

DOCUMENTS (3):
  • Study Protocol (2021-10-27): https://cdn.clinicaltrials.gov/large-docs/68/NCT05141968/Prot_000.pdf
  • Statistical Analysis Plan (2021-10-14): https://cdn.clinicaltrials.gov/large-docs/68/NCT05141968/SAP_001.pdf
  • Informed Consent Form (2017-10-01): https://cdn.clinicaltrials.gov/large-docs/68/NCT05141968/ICF_002.pdf